CLINICAL TRIAL: NCT07360301
Title: Consciousness and Psilocybin Effects on Well-Being: The CoPEWell Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-1861; SMPH | Psychiatry (Other: UW Madison); Protocol Version 12/18/25 (Other: UW Madison)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Well-Being, Psychological; Psychedelic Experiences
MeSH Terms: conditions — Psychological Well-Being | interventions — Psilocybin; Clonidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Psilocybin While Awake, Placebo While Asleep (Experimental): Participants in this group will receive psilocybin by intravenous (IV) infusion while awake and placebo (saline) by IV infusion while asleep during an overnight dosing visit. All participants will also receive oral clonidine prior to dosing to support sleep during the overnight visit.
  Interventions: Drug: Psilocybin; Other: Saline Placebo; Drug: Clonidine
- Placebo While Awake, Psilocybin While Asleep (Experimental): Participants in this group will receive placebo (saline) by intravenous (IV) infusion while awake and psilocybin by IV infusion while asleep during an overnight dosing visit. All participants will also receive oral clonidine prior to dosing to support sleep during the overnight visit.
  Interventions: Drug: Psilocybin; Other: Saline Placebo; Drug: Clonidine
- Placebo While Awake, Placebo While Asleep (Placebo Comparator): Participants in this group will receive placebo (saline) by intravenous (IV) infusion while awake and placebo by IV infusion while asleep during an overnight dosing visit. All participants will also receive oral clonidine prior to dosing to support sleep during the overnight visit.
  Interventions: Other: Saline Placebo; Drug: Clonidine

INTERVENTIONS:
Drug: Psilocybin — IV administration, infusion of 3.2 mg psilocybin over 10 minutes, followed by an additional 0.8 mg infused over the following 20 minutes
  Other Names: intravenous psilocybin
  Arms: Placebo While Awake, Psilocybin While Asleep; Psilocybin While Awake, Placebo While Asleep
Other: Saline Placebo — IV administration, placebo will be 20 mL of saline drawn up aseptically into the same sized (30 mL) syringe as is used for the active drug.
Drug: Clonidine — 0.2 mg of clonidine will be taken by mouth by all participants 60 minutes prior to the initial infusion on Dosing Night
  Other Names: Clonidine ER

SUMMARY:
This study is exploring how psilocybin (a psychedelic drug) may improve mood and wellbeing. Many people report feeling better after taking psilocybin, but it is not clear why. The CoPEWell study will test whether these improvements come from the psychedelic experience itself (the "trip") or from direct effects on the brain. To study this, up to 120 participants will be enrolled to receive psilocybin either while awake or asleep and can expect to be on study for up to 4 months.

DETAILED DESCRIPTION:
Primary Objectives:

1. To evaluate the effect of psilocybin on wellbeing when administered while awake vs. while asleep
2. To evaluate the effect of psilocybin on wellbeing administered while asleep vs. placebo administered while asleep

   Secondary Objectives:
3. To evaluate the effect of psilocybin on psychological flexibility when administered while awake vs. while asleep
4. To evaluate the effect of psilocybin on psychological flexibility administered while asleep vs. placebo administered while asleep
5. To evaluate the effect of psilocybin on social connectedness when administered while awake vs. while asleep
6. To evaluate the effect of psilocybin on social connectedness administered while asleep vs. placebo administered while asleep
7. To evaluate the effect on wellbeing/life satisfaction/purpose/meaning explicitly ascribed to psilocybin administered while awake vs. while asleep
8. To evaluate the effect on wellbeing/life satisfaction/purpose/meaning explicitly ascribed to psilocybin administered while asleep vs. saline placebo administered while asleep

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years (inclusive) at screening, of any identified gender and racial/ethnic group
* Physically healthy; does not meet criteria for an exclusionary medical condition
* No exclusionary sleep condition
* English-speaking (able to provide consent and complete questionnaires)
* Sub-optimal self-reported wellbeing

Exclusion Criteria:

* Exclusionary DSM-5 psychiatric diagnosis and/or active suicidal ideation
* Exclusionary medical conditions or sleep conditions
* Clinically significant safety lab abnormalities (i.e., Complete Blood Count with Differential, Comprehensive Metabolic Panel, and urinalysis)
* Clinically significant electrocardiogram (ECG)
* Use of psychotropic or CNS-altering medications within 3 months of screening
* Hypertension or tachycardia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) score: Psilocybin Awake versus Asleep | Baseline 2 (Day 0) to post-dosing Day 29
  WEMWBS is a 14-item survey scored on a 5 point likert scale. The total range in scores is from 14 to 70 where higher scores indicate better mental wellbeing.
  Reported here for psilocybin administered while awake to psilocybin administered while asleep.
Change in Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) score: Psilocybin Asleep versus Placebo Asleep | Baseline 2 (Day 0) to post-dosing Day 29
  WEMWBS is a 14-item survey scored on a 5 point likert scale. The total range in scores is from 14 to 70 where higher scores indicate better mental wellbeing.
  Reported here for psilocybin administered while asleep to and placebo administered while asleep.

SECONDARY OUTCOMES:
Change in Brief Experiential Avoidance Questionnaire (BEAQ): Psilocybin Awake versus Asleep | Baseline 2 (Day 0) to post-dosing Day 29
  BEAQ is 15-item survey scored on a 6 point likert scale. The total range is scores if from 15 to 90 where higher scores indicating greater avoidance.
  Reported here for psilocybin administered while awake to psilocybin administered while asleep.
Change in Brief Experiential Avoidance Questionnaire (BEAQ): Psilocybin Asleep versus Placebo Asleep | Baseline 2 (Day 0) to post-dosing Day 29
  BEAQ is 15-item survey scored on a 6 point likert scale. The total range is scores if from 15 to 90 where higher scores indicating greater avoidance.
  Reported here for psilocybin administered while asleep to placebo administered while asleep.
Change in Watts Social Connectedness (WCS) Scale: Psilocybin Awake versus Asleep | Baseline 2 (Day 0) to post-dosing Day 29
  WCS is a 19-item survey scored on a visual analog scale. Scores are reported from 0-100 where higher scores interpreted to be more connectedness to others.
  Reported here for psilocybin administered while awake to psilocybin administered while asleep.
Change in Watts Social Connectedness (WCS) Scale: Psilocybin Asleep versus Placebo Asleep | Baseline 2 (Day 0) to post-dosing Day 29
  WCS is a 19-item survey scored on a visual analog scale. Scores are reported from 0-100 where higher scores interpreted to be more connectedness to others.
  Reported here for psilocybin administered while asleep to placebo administered while asleep.
Persisting Effects Questionnaire (PEQ): Psilocybin Awake versus Asleep | post-dosing Day 29
  PEQ-15 is a 15-item survey in which initial items are rated on an 8-point scale ranging from "no more than routine, everyday experiences" to "the single most meaningful experience of my life." Remaining items are rated on a 7-point scale ranging from strong negative change to strong positive change. Higher scores indicate more positive persisting effects.
  Reported here for psilocybin administered while asleep to psilocybin administered while asleep.
Persisting Effects Questionnaire (PEQ): Psilocybin Asleep versus Placebo Asleep | post-dosing Day 29
  PEQ-15 is a 15-item survey in which initial items are rated on an 8-point scale ranging from "no more than routine, everyday experiences" to "the single most meaningful experience of my life." Remaining items are rated on a 7-point scale ranging from strong negative change to strong positive change. Higher scores indicate more positive persisting effects.
  Reported here for psilocybin administered while asleep to psilocybin administered while asleep.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers for research purposes. Data will be shared in accordance with applicable funder requirements, institutional policies, and regulatory obligations, including deposition in a designated data repository when required. Otherwise, data will be shared upon reasonable request following publication of primary study results, subject to institutional review and approval.
Time Frame: Data will be available beginning after publication of primary study results and following completion of data quality control and de-identification procedures.
Access Criteria: Access will be granted to qualified investigators for scientifically valid research proposals, subject to review and approval by the study team and the University of Wisconsin-Madison, and execution of a data use agreement as required.